CLINICAL TRIAL: NCT04327037
Title: Pilot Study of Immunotherapy With ex Vivo Expanded Haploidentical Natural Killer Cells for Leukemia
Brief Title: Safety of Expanded Haploidentical Natural Killer Cells for Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Belarusian Research Center for Pediatric Oncology, Hematology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BelarusianPediatric_NK_Pilot
Record Dates: First submitted 2020-03-18; First posted 2020-03-30 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Leukemia, Acute Myeloid; Leukemia, Acute Lymphoblastic
Keywords: Immunotherapy; Natural killer cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cells + IL-2 (Experimental): After cycle of chemotherapy patient receive one intravenous infusion of expanded haploidentical NK cells on day 0. On alternate days, 6 doses of subcutaneous IL-2 is administered with start on day -1.
  Interventions: Biological: Expanded Haploidentical Natural Killer cells; Drug: IL-2

INTERVENTIONS:
Biological: Expanded Haploidentical Natural Killer cells — One dose (from 20x to >100x 10^6 /kg) of expanded haploidentical NK cells
Drug: IL-2 — 6 doses of IL-2 (1 × 10^6 units/m2) from -1 day every other day.
  Other Names: Ronkoleukinum

SUMMARY:
The purpose of this study is to estimate the safety of ex vivo expanded haploidentical natural killer (NK) cells for patients with leukemia.

DETAILED DESCRIPTION:
Immunotherapy with natural killer (NK) cells may improve the results of treatment for patients with cancer. However, for better efficiency high doses of NK cells are required. For this purpose, NK cells were expanded in the presence of feeder K562 cells gene-modified for expression 4-1BBL and membrane bound IL-21. In the result of expansion, large number of activated NK cells are obtained.

Protocol of immunotherapy includes conditioning (fludarabine + cyclophosphamide or any other protocol of chemotherapy) followed by expanded NK cells intravenous infusion. To sustain proliferation of donor NK cells in vivo patients receive 6 doses of Il-2 every second day. 10 patients will be enrolled in phase I to test different doses of NK cells: 20, 50, 70, 100 and >100 x 10^6/kg.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Relapsed acute myeloid or lymphoblastic leukemia
* Primary refractory myeloid or lymphoblastic leukemia
* Karnofsky or Lansky performance scale greater or equal to 70
* Written informed consent

Donor:

* Haploidentical family donor
* > 18 years old
* Donor suitable for cell donation and apheresis according to standard criteria
* Written informed consent

Exclusion Criteria:

Patients:

* Uncontrolled infection
* Severe hepatic dysfunction: SGOT or SCPT >=5x upper limit of normal for age
* Positive serology for human immunodeficiency virus (HIV)

Donors:

* Pregnancy or breast feeding
* Positive serology for HIV, hepatitis B or C.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 months
  Adverse events will be graded according to the CTCAE v4.0

SECONDARY OUTCOMES:
Days of persistence of adoptively-transferred haploidentical NK cells | 1 months
  Analysis of donor chimerism at +2, 6, 10, 14, 21, 28 days after NK infusion.
Occurrence of disease response | 1 months post infusion
  Analysis of blast cells content in bone marrow by cytomorphology or detection of MRD level by flow/PCR before and after immunotherapy.
Median time to leukocytes and platelets recovery | 2 months post infusion
  Days of platelets (>50x10^9/L) and leukocytes (>1x10^9/L) recovery.
Number of T, B, NK, activated T and NK cells after immunotherapy | 1 months post infusion
  Analysis of T, B, NK, activated T and NK cells numbers (cells/microL) at +2, 6, 10, 14, 21, 28 days after NK infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Aleinikova, Principal Investigator — Belarussian Research Center for Pediatric Oncology, Hematology and Immunology
Locations (1):
- Belarussian Research Center for Pediatric Oncology, Hematology and Immunology, Minsk, Minsk Oblast, Belarus

REFERENCES:
- [Derived] Shman TV, Vashkevich KP, Migas AA, Matveyenka MA, Lasiukov YA, Mukhametshyna NS, Horbach KI, Aleinikova OV. Phenotypic and functional characterisation of locally produced natural killer cells ex vivo expanded with the K562-41BBL-mbIL21 cell line. Clin Exp Med. 2023 Oct;23(6):2551-2560. doi: 10.1007/s10238-022-00974-2. Epub 2022 Dec 17. PMID 36527513